CLINICAL TRIAL: NCT06089512
Title: Comparison of Midpoint Transverse Process to Pleura Block and Thoracic Paravertebral Block for Postoperative Analgesia in Video-Assisted Thoracoscopic Surgery (VATS)"
Brief Title: Comparison of Midpoint Transverse Process to Pleura Block and Thoracic Paravertebral Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Seda Cansabuncu, Principal investigator, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-17/22
Record Dates: First submitted 2023-09-29; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Analgesia; Post Operative Pain
Keywords: thoracic; analgesia; post operative pain; surgery-complication
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): group receiving general anesthesia only
  Interventions: Procedure: Control group
- paravertebral block group (Active Comparator): received single-shot paravertebral block after induction of anesthesia.
  Interventions: Procedure: paravertebral block group
- mid transverse process block group (Active Comparator): received a mid-transverse process -to- pleura block after induction of anesthesia.
  Interventions: Procedure: Mid point transverse process block group

INTERVENTIONS:
Procedure: paravertebral block group — Paravertebral block was applied to the patients after induction of general anesthesia; Intraoperative opioid requirement and postoperative pain scores and analgesic requirement were evaluated.
  Arms: paravertebral block group
Procedure: Mid point transverse process block group — Mid point transverse process block was applied to the patients after induction of general anesthesia; Intraoperative opioid requirement and postoperative pain scores and analgesic requirement were evaluated.
  Arms: mid transverse process block group
Procedure: Control group — Only general anesthesia was applied to the patients.
  Arms: Control group

SUMMARY:
In this study, hypothesis is that the MTPB (mid point transverse process block), which is easier and has fewer complications in patients aged 18-80 undergoing video-assisted thoracic surgery (VATS), provides analgesia as effective as PVB.

DETAILED DESCRIPTION:
Patients between the ages of 18 to 80, scheduled for Video-Assisted Thoracoscopic Surgery (VATS) and classified under the American Society of Anesthesiologists (ASA) class I and II, will be included in the study. Patients with known or suspected local anesthetic allergies, coagulopathy, site injection infections, a history of thoracic surgery, severe neurological or psychiatric disorders, severe cardiovascular diseases, liver failure, kidney failure (glomerular filtration rate <15 ml/min/1.73 m2), and chronic opioid use will be excluded from the study.

Demographic information of the patients (name, protocol number, weight, height, age, body mass index, comorbidities, ASA score) will be recorded. Subsequently, after necessary information is provided, and written and verbal consent is obtained, patients will be randomized into three groups:

Group MTPB: After the induction of general anesthesia and intubation in the operating room, the patient will be placed in the lateral decubitus position. Using ultrasound guidance, a linear probe will be used to perform a MTPB at the midpoint of the superior costotransverse ligament at the level of the 5th intercostal space. A 0.5 ml/kg solution of 0.25% bupivacaine will be administered in-plane.

Group PVB: After the induction of general anesthesia and intubation in the operating room, the patient will be placed in the lateral decubitus position. Using ultrasound guidance, a linear probe will be used to perform a paravertebral block (PVB) at the level of the 5th intercostal space. A 0.5 ml/kg solution of 0.25% bupivacaine will be administered in-plane.

Group P: No peripheral block will be performed in this group.

All patients' hemodynamic data (mean arterial pressure, heart rate, oxygen saturation) will be recorded at 30-minute intervals during the intraoperative period, as well as the amount of opioids used during the surgery. Fifteen minutes before awakening, an intravenous patient-controlled analgesia (PCA) device will be connected, delivering a bolus dose of 2 ml of 1 mg/ml morphine solution with a lockout time of 15 minutes.

During the postoperative period, visual analog pain scores (VAS) will be assessed at 0, 30 minutes, 1, 2, 4, 8, 12, 24, 36, and 48 hours, both at rest and during coughing. Additionally, the time to first analgesic requirement, total analgesic consumption, need for rescue analgesia (contramal 100 mg/2 ml), amount required, possible opioid side effects (nausea, vomiting, respiratory depression, sedation), and time to awakening will be recorded.

The time to first mobilization, postoperative complications, time to discharge, and satisfaction of both patients and the surgical team will be recorded using a 5-point Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 80 years of age
* American Society of Anesthesiologists I-II physical status of and
* Body mass index of 19 to 28 kg/m2

Exclusion Criteria:

* Patients who had coagulopathy
* Previous thoracic surgery
* Emotional instability
* Significant encephalopathy
* Preexisting motor or sensory deficit
* Other contraindications to local anaesthesia, such as allergies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Intraoperative analgesic effects of peripheral blocks | First day
  Investigators will compare the intraoperative analgesic effects by opioid consumption in intraoperative phase.
Postoperative analgesic effects of peripheral blocks | First day
  Visual Analogue Scale (VAS) will be used for postoperative analgesic effects.

SECONDARY OUTCOMES:
opioid consumed through PCA (patient controlled analgesia) | first day
  PCA was used for pain control. An iv solution was prepared to all participants with 100 mg morphine hydrochloride at a concentration of 1 mg/ml in 90 ml saline and the bolus dose was set as 2 ml and the locked time as 15 min. From the recovery unit, a bolus dose of morphine was administered with the PCA device if VAS≥4 by questioning or upon the request of the participants. Participants who had VAS≥4 despite PCA were administered 50 mg dexketoprofen iv as rescue analgesic and 50 mg tramadol intramuscularly as the second rescue analgesic if VAS≥4 continued.
Side effects | First day
  The necessity for supplementary analgesics, any complications associated with the puncture procedure such as infection, hematoma, and pneumothorax (confirmed via direct thoracoscopic visualization), the incidence of postoperative nausea and vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: seda cansabuncu, Principal Investigator — BURSA ULUDAG UNIVERSITY HOSPITAL
Locations (1):
- Bursa Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
we plan share ,study Protocol, statistical Analysis Plan (SAP), informed Consent Form (ICF)